CLINICAL TRIAL: NCT01422876
Title: A Phase III Randomized, Double-blind, Parallel Group Study to Evaluate the Efficacy and Safety of Once Daily Oral Administration of BI 10773 25 mg/Linagliptin 5 mg and BI 10773 10 mg/Linagliptin 5 mg Fixed Dose Combination Tablets Compared With the Individual Components (BI 10773 25 mg, BI 10773 10 mg, and Linagliptin 5 mg) for 52 Weeks in Treatment naïve and Metformin Treated Patients With Type 2 Diabetes Mellitus With Insufficient Glycaemic Control
Brief Title: Efficacy and Safety of Empagliflozin (BI 10773) / Linagliptin (BI 1356) Fixed Dose Combination in Treatment naïve and Metformin Treated Type 2 Diabetes Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1275.1; 2011-000383-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Linagliptin

ARMS (5):
- BI 10773/linagliptin FDC (high dose) (Experimental): Patients receive BI 10773/linagliptin FDC (high dose) once daily
  Interventions: Drug: high dose FDC; Drug: low dose FDC placebo; Drug: high dose BI 10773 placebo; Drug: BI 10773 low dose placebo; Drug: linagliptin placebo
- BI 10773/linagliptin FDC (low dose) (Experimental): Patients receive BI 10773/linagliptin FDC (low dose) once daily
  Interventions: Drug: high dose FDC placebo; Drug: low dose FDC; Drug: high dose BI 10773 placebo; Drug: BI 10773 low dose placebo; Drug: linagliptin placebo
- BI 10773 (high dose) (Active Comparator): Patients receive BI 10773 (high dose) once daily
  Interventions: Drug: BI 10773 high dose; Drug: high dose FDC placebo; Drug: low dose FDC placebo; Drug: low dose BI 10773 placebo; Drug: linagliptin placebo
- BI 10773 (low dose) (Active Comparator): Patients receive BI 10773 (low dose) once daily
  Interventions: Drug: high dose FDC placebo; Drug: low dose FDC placebo; Drug: high dose BI 10773 placebo; Drug: BI 10773 low dose; Drug: linagliptin placebo
- Linagliptin (Active Comparator): Patients receive linagliptin once daily
  Interventions: Drug: low dose FDC placebo; Drug: high dose FDC placebo; Drug: linagliptin; Drug: high dose BI 10773 placebo; Drug: low dose BI 10773 placebo

INTERVENTIONS:
Drug: high dose FDC — once daily
  Arms: BI 10773/linagliptin FDC (high dose)
Drug: BI 10773 high dose — once daily
  Arms: BI 10773 (high dose)
Drug: high dose FDC placebo — once daily
  Arms: BI 10773 (low dose)
Drug: low dose FDC placebo — once daily
  Arms: BI 10773/linagliptin FDC (high dose)
Drug: high dose FDC placebo — once daily
  Arms: BI 10773/linagliptin FDC (low dose)
Drug: high dose FDC placebo — once daily
  Arms: BI 10773 (high dose)
Drug: low dose FDC placebo — once daily
  Arms: BI 10773 (low dose)
Drug: low dose FDC placebo — once daily
  Arms: Linagliptin
Drug: high dose BI 10773 placebo — once daily
  Arms: BI 10773 (low dose)
Drug: low dose FDC — once daily
  Arms: BI 10773/linagliptin FDC (low dose)
Drug: high dose FDC placebo — once daily
  Arms: Linagliptin
Drug: BI 10773 low dose — low dose once daily
  Arms: BI 10773 (low dose)
Drug: high dose BI 10773 placebo — once daily
  Arms: BI 10773/linagliptin FDC (high dose)
Drug: high dose BI 10773 placebo — once daily
  Arms: BI 10773/linagliptin FDC (low dose)
Drug: linagliptin — once daily
  Arms: Linagliptin
Drug: low dose FDC placebo — once daily
  Arms: BI 10773 (high dose)
Drug: linagliptin placebo — once daily
  Arms: BI 10773 (low dose)
Drug: BI 10773 low dose placebo — once daily
  Arms: BI 10773/linagliptin FDC (high dose)
Drug: linagliptin placebo — once daily
  Arms: BI 10773/linagliptin FDC (high dose)
Drug: low dose BI 10773 placebo — once daily
  Arms: BI 10773 (high dose)
Drug: linagliptin placebo — once daily
  Arms: BI 10773 (high dose)
Drug: high dose BI 10773 placebo — once daily
  Arms: Linagliptin
Drug: BI 10773 low dose placebo — once daily
  Arms: BI 10773/linagliptin FDC (low dose)
Drug: low dose BI 10773 placebo — once daily
  Arms: Linagliptin
Drug: linagliptin placebo — once daily
  Arms: BI 10773/linagliptin FDC (low dose)

SUMMARY:
This trial will evaluate use of BI 10773/linagliptin once daily (qd) fixed dose combination (FDC) in treatment naïve and metformin treated patients with type 2 diabetes mellitus to support approval by regulatory authorities.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of type 2 diabetes mellitus prior to informed consent
2. Male and female patients on diet and exercise regimen who are drug-naïve (defined as absence of any oral antidiabetic therapy, glucagon like peptide-1 analog or insulin for 12 weeks prior to randomization) or pre-treated with metformin (=1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation.
3. Glycosylated hemoglobin (HbA1c) = 7.0% and = 10.5% (= 53.0 mmol/mol and = 91.3 mmol/mol) at Visit 1 (screening)

Exclusion criteria:

1. Uncontrolled hyperglycemia with a glucose level >240 mg/dl (>13.3 mmol/L) after an overnight fast during placebo run-in and confirmed by a second measurement (not on the same day).
2. Any other antidiabetic drug within 12 weeks prior to randomization (except metformin background therapy as defined via inclusion criterion 2)
3. Acute coronary syndrome (non-ST elevation myocardial infarction, ST elevation myocardial infarction and unstable angina pectoris), stroke or (transient ischemic attack) TIA within 3 months prior to informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1405 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (211):
- United States (112):
  - 1275.1.01103 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1275.1.01107 Boehringer Ingelheim Investigational Site, Foley, Alabama
  - 1275.1.01043 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1275.1.01066 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1275.1.01047 Boehringer Ingelheim Investigational Site, Pell City, Alabama
  - 1275.1.01089 Boehringer Ingelheim Investigational Site, Mesa, Arizona
  - 1275.1.01064 Boehringer Ingelheim Investigational Site, Tempe, Arizona
  - 1275.1.01028 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1275.1.01086 Boehringer Ingelheim Investigational Site, Cerritos, California
  - 1275.1.01067 Boehringer Ingelheim Investigational Site, Chula Vista, California
  - 1275.1.01109 Boehringer Ingelheim Investigational Site, Encino, California
  - 1275.1.01012 Boehringer Ingelheim Investigational Site, Fresno, California
  - 1275.1.01050 Boehringer Ingelheim Investigational Site, Harbor City, California
  - 1275.1.01056 Boehringer Ingelheim Investigational Site, Huntington Park, California
  - 1275.1.01021 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1275.1.01024 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1275.1.01112 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1275.1.01083 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 1275.1.01071 Boehringer Ingelheim Investigational Site, San Dimas, California
  - 1275.1.01044 Boehringer Ingelheim Investigational Site, Tustin, California
  - 1275.1.01078 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1275.1.01124 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1275.1.01010 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1275.1.01048 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1275.1.01073 Boehringer Ingelheim Investigational Site, Gainesville, Florida
  - 1275.1.01063 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1275.1.01077 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1275.1.01090 Boehringer Ingelheim Investigational Site, Inverness, Florida
  - 1275.1.01054 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1275.1.01092 Boehringer Ingelheim Investigational Site, Maitland, Florida
  - 1275.1.01065 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1275.1.01110 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1275.1.01040 Boehringer Ingelheim Investigational Site, Miami Beach, Florida
  - 1275.1.01025 Boehringer Ingelheim Investigational Site, Miami Lakes, Florida
  - 1275.1.01094 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1275.1.01068 Boehringer Ingelheim Investigational Site, Ormond Beach, Florida
  - 1275.1.01051 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1275.1.01079 Boehringer Ingelheim Investigational Site, Port Orange, Florida
  - 1275.1.01117 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1275.1.01039 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1275.1.01007 Boehringer Ingelheim Investigational Site, Marietta, Georgia
  - 1275.1.01111 Boehringer Ingelheim Investigational Site, Norcross, Georgia
  - 1275.1.01076 Boehringer Ingelheim Investigational Site, Savannah, Georgia
  - 1275.1.01100 Boehringer Ingelheim Investigational Site, Addison, Illinois
  - 1275.1.01042 Boehringer Ingelheim Investigational Site, Des Moines, Iowa
  - 1275.1.01059 Boehringer Ingelheim Investigational Site, Paducah, Kentucky
  - 1275.1.01003 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 1275.1.01125 Boehringer Ingelheim Investigational Site, Hyattsville, Maryland
  - 1275.1.01081 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1275.1.01085 Boehringer Ingelheim Investigational Site, Rochester, Michigan
  - 1275.1.01035 Boehringer Ingelheim Investigational Site, Southfield, Michigan
  - 1275.1.01023 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1275.1.01027 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1275.1.01033 Boehringer Ingelheim Investigational Site, Great Falls, Montana
  - 1275.1.01099 Boehringer Ingelheim Investigational Site, Henderson, Nevada
  - 1275.1.01101 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1275.1.01114 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1275.1.01123 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1275.1.01013 Boehringer Ingelheim Investigational Site, Elizabeth, New Jersey
  - 1275.1.01057 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1275.1.01002 Boehringer Ingelheim Investigational Site, Binghamton, New York
  - 1275.1.01020 Boehringer Ingelheim Investigational Site, Endwell, New York
  - 1275.1.01095 Boehringer Ingelheim Investigational Site, Flushing, New York
  - 1275.1.01062 Boehringer Ingelheim Investigational Site, Glens Falls, New York
  - 1275.1.01006 Boehringer Ingelheim Investigational Site, New York, New York
  - 1275.1.01011 Boehringer Ingelheim Investigational Site, Asheboro, North Carolina
  - 1275.1.01052 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 1275.1.01045 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1275.1.01001 Boehringer Ingelheim Investigational Site, Akron, Ohio
  - 1275.1.01032 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1275.1.01061 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1275.1.01116 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1275.1.01016 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1275.1.01102 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1275.1.01017 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1275.1.01036 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1275.1.01030 Boehringer Ingelheim Investigational Site, Delaware, Ohio
  - 1275.1.01055 Boehringer Ingelheim Investigational Site, Groveport, Ohio
  - 1275.1.01075 Boehringer Ingelheim Investigational Site, Wadsworth, Ohio
  - 1275.1.01034 Boehringer Ingelheim Investigational Site, Norman, Oklahoma
  - 1275.1.01082 Boehringer Ingelheim Investigational Site, Corvallis, Oregon
  - 1275.1.01084 Boehringer Ingelheim Investigational Site, Altoona, Pennsylvania
  - 1275.1.01038 Boehringer Ingelheim Investigational Site, Fleetwood, Pennsylvania
  - 1275.1.01019 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1275.1.01072 Boehringer Ingelheim Investigational Site, Scottdale, Pennsylvania
  - 1275.1.01088 Boehringer Ingelheim Investigational Site, Tipton, Pennsylvania
  - 1275.1.01014 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 1275.1.01060 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 1275.1.01093 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1275.1.01122 Boehringer Ingelheim Investigational Site, Florence, South Carolina
  - 1275.1.01005 Boehringer Ingelheim Investigational Site, Hodges, South Carolina
  - 1275.1.01015 Boehringer Ingelheim Investigational Site, Brentwood, Tennessee
  - 1275.1.01031 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 1275.1.01121 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1275.1.01069 Boehringer Ingelheim Investigational Site, Spring Hill, Tennessee
  - 1275.1.01049 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1275.1.01080 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1275.1.01029 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1275.1.01053 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1275.1.01106 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1275.1.01018 Boehringer Ingelheim Investigational Site, Pearland, Texas
  - 1275.1.01096 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1275.1.01113 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1275.1.01120 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1275.1.01105 Boehringer Ingelheim Investigational Site, Spring, Texas
  - 1275.1.01037 Boehringer Ingelheim Investigational Site, Waco, Texas
  - 1275.1.01008 Boehringer Ingelheim Investigational Site, Bountiful, Utah
  - 1275.1.01022 Boehringer Ingelheim Investigational Site, West Jordan, Utah
  - 1275.1.01091 Boehringer Ingelheim Investigational Site, South Chesterfield, Virginia
  - 1275.1.01118 Boehringer Ingelheim Investigational Site, Selah, Washington
  - 1275.1.01087 Boehringer Ingelheim Investigational Site, Shoreline, Washington
  - 1275.1.01119 Boehringer Ingelheim Investigational Site, Spokane, Washington
- Argentina (5):
  - 1275.1.54001 Boehringer Ingelheim Investigational Site, Caba
  - 1275.1.54005 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1275.1.54003 Boehringer Ingelheim Investigational Site, Córdoba
  - 1275.1.54004 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1275.1.54002 Boehringer Ingelheim Investigational Site, Mendoza
- Australia (2):
  - 1275.1.61003 Boehringer Ingelheim Investigational Site, Wollongong, New South Wales
  - 1275.1.61002 Boehringer Ingelheim Investigational Site, East Ringwood, Victoria
- Brazil (3):
  - 1275.1.55002 Boehringer Ingelheim Investigational Site, Joaquim Távora
  - 1275.1.55001 Boehringer Ingelheim Investigational Site, Rio de Janeiro - RJ
  - 1275.1.55005 Boehringer Ingelheim Investigational Site, São Paulo
- Bulgaria (3):
  - 1275.1.59003 Boehringer Ingelheim Investigational Site, Plovdiv
  - 1275.1.59006 Boehringer Ingelheim Investigational Site, Rousse
  - 1275.1.59004 Boehringer Ingelheim Investigational Site, Sofia
- Canada (8):
  - 1275.1.20008 Boehringer Ingelheim Investigational Site, Bathurst, New Brunswick
  - 1275.1.20007 Boehringer Ingelheim Investigational Site, Bay Roberts, Newfoundland and Labrador
  - 1275.1.20006 Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - 1275.1.20004 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1275.1.20001 Boehringer Ingelheim Investigational Site, Brampton, Ontario
  - 1275.1.20005 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1275.1.20003 Boehringer Ingelheim Investigational Site, Drummondville, Quebec
  - 1275.1.20002 Boehringer Ingelheim Investigational Site, Pointe-Claire, Quebec
- Colombia (4):
  - 1275.1.57004 Boehringer Ingelheim Investigational Site, Barranquilla
  - 1275.1.57002 Boehringer Ingelheim Investigational Site, Bogotá
  - 1275.1.57005 Boehringer Ingelheim Investigational Site, Bogotá
  - 1275.1.57003 Boehringer Ingelheim Investigational Site, Tolima
- Denmark (3):
  - 1275.1.45004 Boehringer Ingelheim Investigational Site, Aalborg
  - 1275.1.45003 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1275.1.45002 Boehringer Ingelheim Investigational Site, København NV
- Estonia (5):
  - 1275.1.37206 Boehringer Ingelheim Investigational Site, Kiviõli
  - 1275.1.37202 Boehringer Ingelheim Investigational Site, Pärnu
  - 1275.1.37201 Boehringer Ingelheim Investigational Site, Tallinn
  - 1275.1.37204 Boehringer Ingelheim Investigational Site, Tallinn
  - 1275.1.37203 Boehringer Ingelheim Investigational Site, Viljandi County
- Hungary (3):
  - 1275.1.36002 Boehringer Ingelheim Investigational Site, Budapest
  - 1275.1.36003 Boehringer Ingelheim Investigational Site, Budapest
  - 1275.1.36001 Boehringer Ingelheim Investigational Site, Gyöngyös
- Italy (4):
  - 1275.1.39003 Boehringer Ingelheim Investigational Site, Bassano Del Grappa (VI)
  - 1275.1.39002 Boehringer Ingelheim Investigational Site, Fermo
  - 1275.1.39001 Boehringer Ingelheim Investigational Site, Milan
  - 1275.1.39004 Boehringer Ingelheim Investigational Site, Roma
- Lebanon (6):
  - 1275.1.96004 Boehringer Ingelheim Investigational Site, Baabda
  - 1275.1.96002 Boehringer Ingelheim Investigational Site, Beirut
  - 1275.1.96003 Boehringer Ingelheim Investigational Site, Beirut
  - 1275.1.96006 Boehringer Ingelheim Investigational Site, Beirut
  - 1275.1.96008 Boehringer Ingelheim Investigational Site, Beirut
  - 1275.1.96007 Boehringer Ingelheim Investigational Site, Saida
- Malaysia (2):
  - 1275.1.60001 Boehringer Ingelheim Investigational Site, Kedah
  - 1275.1.60002 Boehringer Ingelheim Investigational Site, Perak
- Mexico (5):
  - 1275.1.52002 Boehringer Ingelheim Investigational Site, México
  - 1275.1.52005 Boehringer Ingelheim Investigational Site, México
  - 1275.1.52003 Boehringer Ingelheim Investigational Site, Monterrey
  - 1275.1.52001 Boehringer Ingelheim Investigational Site, Pachuca
  - 1275.1.52004 Boehringer Ingelheim Investigational Site, San Luis Potosí City
- Peru (5):
  - 1275.1.51001 Boehringer Ingelheim Investigational Site, Arequipa
  - 1275.1.51003 Boehringer Ingelheim Investigational Site, Ica
  - 1275.1.51002 Boehringer Ingelheim Investigational Site, Lima
  - 1275.1.51004 Boehringer Ingelheim Investigational Site, Lima
  - 1275.1.51005 Boehringer Ingelheim Investigational Site, Lima
- Philippines (6):
  - 1275.1.63002 Boehringer Ingelheim Investigational Site, Davao City
  - 1275.1.63001 Boehringer Ingelheim Investigational Site, Greenhills, San Juan
  - 1275.1.63004 Boehringer Ingelheim Investigational Site, Manila
  - 1275.1.63006 Boehringer Ingelheim Investigational Site, Marikina City
  - 1275.1.63003 Boehringer Ingelheim Investigational Site, Pasay
  - 1275.1.63005 Boehringer Ingelheim Investigational Site, Pasig
- Poland (4):
  - 1275.1.48002 Boehringer Ingelheim Investigational Site, Lodz
  - 1275.1.48004 Boehringer Ingelheim Investigational Site, Poznan
  - 1275.1.48001 Boehringer Ingelheim Investigational Site, Warsaw
  - 1275.1.48003 Boehringer Ingelheim Investigational Site, Warsaw
- Romania (10):
  - 1275.1.40001 Boehringer Ingelheim Investigational Site, Alba Iulia
  - 1275.1.40005 Boehringer Ingelheim Investigational Site, Baia Mare Maramures
  - 1275.1.40004 Boehringer Ingelheim Investigational Site, Brasov
  - 1275.1.40008 Boehringer Ingelheim Investigational Site, Bucharest
  - 1275.1.40009 Boehringer Ingelheim Investigational Site, Bucharest
  - 1275.1.40006 Boehringer Ingelheim Investigational Site, Cluj-Napoca
  - 1275.1.40007 Boehringer Ingelheim Investigational Site, Galati
  - 1275.1.40002 Boehringer Ingelheim Investigational Site, Oradea
  - 1275.1.40010 Boehringer Ingelheim Investigational Site, Sibiu
  - 1275.1.40003 Boehringer Ingelheim Investigational Site, Târgu Mureş
- Russia (6):
  - 1275.1.70006 Boehringer Ingelheim Investigational Site, Arkhangelsk
  - 1275.1.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 1275.1.70002 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1275.1.70003 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1275.1.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1275.1.70004 Boehringer Ingelheim Investigational Site, Samara
- Spain (5):
  - 1275.1.34004 Boehringer Ingelheim Investigational Site, Barcelona
  - 1275.1.34005 Boehringer Ingelheim Investigational Site, Barcelona
  - 1275.1.34002 Boehringer Ingelheim Investigational Site, Hospitalet de Llobegrat
  - 1275.1.34003 Boehringer Ingelheim Investigational Site, Palma de Mallorca
  - 1275.1.34006 Boehringer Ingelheim Investigational Site, Tarragona
- Sweden (3):
  - 1275.1.46003 Boehringer Ingelheim Investigational Site, Järfälla
  - 1275.1.46004 Boehringer Ingelheim Investigational Site, Rättvik
  - 1275.1.46002 Boehringer Ingelheim Investigational Site, Skene
- Taiwan (7):
  - 1275.1.88006 Chang Gung Memorial Hospital-CY, Chiayi City
  - 1275.1.88007 E-Da Hospital, Kaohsiung City
  - 1275.1.88001 Cardinal Tien Hospital, New Taipei City
  - 1275.1.88004 Taichung Veterans General Hospital, Taichung
  - 1275.1.88008 Chi Mei Medical Center, Tainan
  - 1275.1.88002 Far Eastern Memorial Hospital, Taipei
  - 1275.1.88003 Taipei Chang Gung Memorial Hospital, Taipei

REFERENCES:
- [Derived] DeFronzo RA, Lee C, Kohler S. Safety and Tolerability of Combinations of Empagliflozin and Linagliptin in Patients with Type 2 Diabetes: Pooled Data from Two Randomized Controlled Trials. Adv Ther. 2018 Jul;35(7):1009-1022. doi: 10.1007/s12325-018-0724-y. Epub 2018 Jun 15. PMID 29949041
- [Derived] Lewin A, DeFronzo RA, Patel S, Liu D, Kaste R, Woerle HJ, Broedl UC. Initial combination of empagliflozin and linagliptin in subjects with type 2 diabetes. Diabetes Care. 2015 Mar;38(3):394-402. doi: 10.2337/dc14-2365. Epub 2015 Jan 29. PMID 25633662
- [Derived] DeFronzo RA, Lewin A, Patel S, Liu D, Kaste R, Woerle HJ, Broedl UC. Combination of empagliflozin and linagliptin as second-line therapy in subjects with type 2 diabetes inadequately controlled on metformin. Diabetes Care. 2015 Mar;38(3):384-93. doi: 10.2337/dc14-2364. Epub 2015 Jan 12. PMID 25583754

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1405 patients enrolled and randomized the data for 42 randomized patients were excluded from all analyses due to serious non-compliance. Therefore, 1363 patients were included in the analyses.
Groups:
- Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation. Test product: Empagliflozin/linagliptin FDC tablets dose: 25 mg/5 mg q.d. mode of admin: Oral
- Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation.
  Test product: Empagliflozin/linagliptin FDC tablets dose: 10 mg/5 mg q.d. mode of admin.: Oral
- Metformin Background: Empagliflozin 25 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation.
  Reference therapy 1: Empagliflozin tablets dose: 25 mg q.d. mode of admin.: Oral
- Metformin Background: Empagliflozin 10 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation.
  Reference therapy 1: Empagliflozin tablets dose: 10 mg q.d. mode of admin.: Oral
- Metformin Background: Linagliptin 5 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation.
  Reference therapy 2: Linagliptin tablets dose: 5 mg q.d. mode of admin.: Oral
- Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg: Study population treatment naive defined as an absence of any oral antidiabetic therapy, GLP-1 analog or insulin for 12 weeks prior to randomisation.
  Test product: Empagliflozin/linagliptin FDC tablets dose: 25 mg/5 mg q.d. mode of admin.: Oral
- Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg: Study population treatment naive defined as an absence of any oral antidiabetic therapy, GLP-1 analog or insulin for 12 weeks prior to randomisation.
  Test product: Empagliflozin/linagliptin FDC tablets dose: 10 mg/5 mg q.d. mode of admin.: Oral
- Treatment Naive: Empagliflozin 25 mg: Study population treatment naive defined as an absence of any oral antidiabetic therapy, GLP-1 analog or insulin for 12 weeks prior to randomisation.
  Reference therapy 1: Empagliflozin tablets dose: 25 mg q.d. mode of admin.: Oral
- Treatment Naive: Empagliflozin 10 mg: Study population treatment naive defined as an absence of any oral antidiabetic therapy, GLP-1 analog or insulin for 12 weeks prior to randomisation.
  Reference therapy 1: Empagliflozin tablets dose: 10 mg q.d. mode of admin.: Oral
- Treatment Naive: Linagliptin 5 mg: Study population treatment naive defined as an absence of any oral antidiabetic therapy, GLP-1 analog or insulin for 12 weeks prior to randomisation.
  Reference therapy 2: Linagliptin tablets dose: 5 mg q.d. mode of admin.: Oral
Period: Week 24
Arm/Group | Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 25 mg | Metformin Background: Empagliflozin 10 mg | Metformin Background: Linagliptin 5 mg | Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg | Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg | Treatment Naive: Empagliflozin 25 mg | Treatment Naive: Empagliflozin 10 mg | Treatment Naive: Linagliptin 5 mg
Started | 137 | 136 | 141 | 140 | 132 | 137 | 136 | 135 | 134 | 135
Completed | 131 | 133 | 136 | 132 | 125 | 131 | 130 | 128 | 128 | 125
Not Completed | 6 | 3 | 5 | 8 | 7 | 6 | 6 | 7 | 6 | 10
Not completed — Lost to Follow-up | 1 | 1 | 2 | 4 | 2 | 0 | 1 | 3 | 3 | 4
Not completed — Consent withdrawn | 5 | 1 | 3 | 4 | 5 | 6 | 5 | 4 | 3 | 6
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 52
Arm/Group | Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 25 mg | Metformin Background: Empagliflozin 10 mg | Metformin Background: Linagliptin 5 mg | Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg | Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg | Treatment Naive: Empagliflozin 25 mg | Treatment Naive: Empagliflozin 10 mg | Treatment Naive: Linagliptin 5 mg
Started | 137 | 136 | 141 | 140 | 132 | 137 | 136 | 135 | 134 | 135
Completed | 125 | 126 | 128 | 122 | 117 | 120 | 120 | 112 | 113 | 118
Not Completed | 12 | 10 | 13 | 18 | 15 | 17 | 16 | 23 | 21 | 17
Not completed — Lost to Follow-up | 3 | 5 | 7 | 5 | 8 | 5 | 5 | 8 | 7 | 8
Not completed — Consent withdrawn | 9 | 4 | 6 | 12 | 7 | 12 | 10 | 12 | 13 | 9
Not completed — Death | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: FAS
Groups:
- Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation and treatment naive defined as an absence of any oral antidiabetic therapy, GLP-1 analog or insulin for 12 weeks prior to randomisation.
  . Test product: Empagliflozin/linagliptin FDC tablets dose: 25 mg/5 mg q.d. mode of admin.: Oral
- Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation and treatment naive defined as an absence of any oral antidiabetic therapy, GLP-1 analog or insulin for 12 weeks prior to randomisation.
  Test product: Empagliflozin/linagliptin FDC tablets dose: 10 mg/5 mg q.d. mode of admin.: Oral
- Metformin Background: Empagliflozin 25 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation and treatment naive defined as an absence of any oral antidiabetic therapy, GLP-1 analog or insulin for 12 weeks prior to randomisation.
  Reference therapy 1: Empagliflozin tablets dose: 25 mg q.d. mode of admin.: Oral
- Metformin Background: Empagliflozin 10 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation and treatment naive defined as an absence of any oral antidiabetic therapy, GLP-1 analog or insulin for 12 weeks prior to randomisation.
  Reference therapy 1: Empagliflozin tablets dose: 10 mg q.d. mode of admin.: Oral
- Metformin Background: Linagliptin 5 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation and treatment naive defined as an absence of any oral antidiabetic therapy, GLP-1 analog or insulin for 12 weeks prior to randomisation.
  Reference therapy 2: Linagliptin tablets dose: 5 mg q.d. mode of admin.: Oral
- Total: Total of all reporting groups
Arm/Group | Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 25 mg | Metformin Background: Empagliflozin 10 mg | Metformin Background: Linagliptin 5 mg | Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg | Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg | Treatment Naive: Empagliflozin 25 mg | Treatment Naive: Empagliflozin 10 mg | Treatment Naive: Linagliptin 5 mg | Total
Number analyzed (Participants) | 134 | 135 | 140 | 137 | 128 | 134 | 135 | 133 | 132 | 133 | 1341
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.2) | 56.2 (10.3) | 55.5 (10.0) | 56.1 (10.5) | 56.2 (10.0) | 54.2 (10.0) | 55.2 (9.8) | 56.0 (9.3) | 53.9 (10.5) | 53.8 (11.5) | 55.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 52 | 75 | 59 | 64 | 64 | 62 | 56 | 68 | 58 | 620
  Male | 72 | 83 | 65 | 78 | 64 | 70 | 73 | 77 | 64 | 75 | 721

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) for Metformin Background Patients
Description: Glycosylated hemoglobin (HbA1c) is a measurement of the percentage of hemoglobin that is glycated. The change from baseline in HbA1c is calculated as the week 24 HbA1c minus the baseline HbA1c. Since HbA1c is measured as a percentage the change from baseline is also a percentage.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF). FAS - all Metformin Background patients randomised and treated who had a baseline and at least 1 on treatment HbA1c value.
Measure: Least Squares Mean (Standard Error); unit: % change from baseline
Groups:
- Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation.
  Test product: Empagliflozin/linagliptin FDC tablets dose: 25 mg/5 mg q.d. mode of admin.: Oral
Arm/Group | Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 25 mg | Metformin Background: Empagliflozin 10 mg | Metformin Background: Linagliptin 5 mg
Number analyzed (Participants) | 134 | 135 | 140 | 137 | 128
% change from baseline | -1.19 (0.06) | -1.08 (0.06) | -0.62 (0.06) | -0.66 (0.06) | -0.70 (0.06)
Statistical Analysis 1: Comparison: Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg vs Metformin Background: Empagliflozin 25 mg; Model for Week 24 includes baseline HbA1c (p<0.0001) as linear covariate(s) and baseline eGFR (MDRD) (p=0.0038), geographical region (p<0.0001), treatment (p<0.0001) as fixed effect(s); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.58, 95% CI 2-sided [-0.75 to -0.41], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg vs Metformin Background: Linagliptin 5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.50, 95% CI 2-sided [-0.67 to -0.32], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg vs Metformin Background: Empagliflozin 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.59 to -0.25], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg vs Metformin Background: Linagliptin 5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.39, 95% CI 2-sided [-0.56 to -0.21], Standard Error of Mean 0.09

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 24 for Metformin Background Patients
Description: Change from baseline in fasting plasma glucose at week 24 for Metformin Background patients.
Time Frame: Baseline and 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL change from baseline
Groups:
- Metformin Background: Empagliflozin 10 mg: Study population on a stable background of metformin defined as pre-treated with metformin (≥1500 mg/day or on the maximum tolerated dose or the maximum dose according to local label) unchanged for 12 weeks prior to randomisation.
  Reference therapy 1: Empagliflozin tablets dose: 10 mg q.d. mode of admin.: Ora
Arm/Group | Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 25 mg | Metformin Background: Empagliflozin 10 mg | Metformin Background: Linagliptin 5 mg
Number analyzed (Participants) | 133 | 134 | 139 | 136 | 127
mg/dL change from baseline | -35.25 (2.53) | -32.18 (2.52) | -18.83 (2.47) | -20.84 (2.50) | -13.05 (2.59)
Statistical Analysis 1: Comparison: Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg vs Metformin Background: Empagliflozin 25 mg; Model for Week 24 includes baseline fasting plasma glucose (p<0.0001), baseline HbA1c (p=0.6082) as linear covariate(s) and baseline eGFR (MDRD) (p=0.3685), geographical region (p=0.0104), treatment (p<0.0001) as fixed effect(s); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -16.43, 95% CI 2-sided [-23.37 to -9.48], Standard Error of Mean 3.54
Statistical Analysis 2: Comparison: Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg vs Metformin Background: Linagliptin 5 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -22.20, 95% CI 2-sided [-29.30 to -15.10], Standard Error of Mean 3.62
Statistical Analysis 3: Comparison: Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg vs Metformin Background: Empagliflozin 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0015, ANCOVA; Mean Difference (Net) = -11.34, 95% CI 2-sided [-18.31 to -4.37], Standard Error of Mean 3.55
Statistical Analysis 4: Comparison: Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg vs Metformin Background: Linagliptin 5 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -19.12, 95% CI 2-sided [-26.21 to -12.03], Standard Error of Mean 3.61

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 24 for Treatment Naive Patients
Description: Change from baseline in fasting plasma glucose at week 24 for Treatment Naive patients.
Time Frame: Baseline and 24 Weeks
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF). FAS - all treatment naive patients randomised and treated who had a baseline and at least 1 on treatment HbA1c value.
Measure: Least Squares Mean (Standard Error); unit: mg/dL change from baseline
Arm/Group | Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg | Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg | Treatment Naive: Empagliflozin 25 mg | Treatment Naive: Empagliflozin 10 mg | Treatment Naive: Linagliptin 5 mg
Number analyzed (Participants) | 134 | 135 | 133 | 132 | 133
mg/dL change from baseline | -29.55 (2.67) | -28.21 (2.66) | -24.24 (2.68) | -22.39 (2.69) | -5.92 (2.68)
Statistical Analysis 1: Comparison: Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg vs Treatment Naive: Empagliflozin 25 mg; Model for Week 24 includes baseline fasting plasma glucose (p<0.0001), baseline HbA1c (p=0.4591) as linear covariate(s) and baseline eGFR (MDRD) (p=0.7413), geographical region (p=0.1504), treatment (p<0.0001) as fixed effect(s); Test type: Superiority or Other; p = 0.1605, ANCOVA; Mean Difference (Net) = -5.31, 95% CI 2-sided [-12.74 to 2.11], Standard Error of Mean 3.78
Statistical Analysis 2: Comparison: Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg vs Treatment Naive: Empagliflozin 10 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1246, ANCOVA; Mean Difference (Net) = -5.82, 95% CI 2-sided [-13.25 to 1.61], Standard Error of Mean 3.78
Statistical Analysis 3: Comparison: Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg vs Treatment Naive: Linagliptin 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -23.63, 95% CI 2-sided [-31.06 to -16.21], Standard Error of Mean 3.78
Statistical Analysis 4: Comparison: Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg vs Treatment Naive: Linagliptin 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -22.29, 95% CI 2-sided [-29.71 to -14.88], Standard Error of Mean 3.77

4. Secondary Outcome: Change From Baseline in Body Weight for Metformin Background Patients
Description: Change from baseline in body weight for Metformin Background patients.
Time Frame: Baseline and 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg change from baseline
Arm/Group | Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 25 mg | Metformin Background: Empagliflozin 10 mg | Metformin Background: Linagliptin 5 mg
Number analyzed (Participants) | 134 | 135 | 140 | 137 | 128
kg change from baseline | -2.99 (0.31) | -2.60 (0.30) | -3.18 (0.30) | -2.53 (0.30) | -0.69 (0.31)
Statistical Analysis 1: Comparison: Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg vs Metformin Background: Empagliflozin 25 mg; Model for Week 24 includes baseline weight (p<0.0001), baseline HbA1c (p=0.1610) as linear covariate(s) and baseline eGFR (MDRD) (p=0.3685), geographical region (p=0.0162), treatment (p<0.0001) as fixed effect(s); Test type: Superiority or Other; p = 0.6604, ANCOVA — Not an alpha protected test; Mean Difference (Net) = 0.19, 95% CI 2-sided [-0.65 to 1.03], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg vs Metformin Background: Linagliptin 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -2.30, 95% CI 2-sided [-3.15 to -1.44], Standard Error of Mean 0.44
Statistical Analysis 3: Comparison: Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg vs Metformin Background: Empagliflozin 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.8757, ANCOVA — Not an alpha protected test; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.91 to 0.77], Standard Error of Mean 0.43
Statistical Analysis 4: Comparison: Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg vs Metformin Background: Linagliptin 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -1.91, 95% CI 2-sided [-2.77 to -1.05], Standard Error of Mean 0.44

5. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) for Treatment Naive Patients
Description: as for outcome 1
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF). FAS - all treatment naive patients randomised to and treated who had a baseline and at least 1 on treatment HbA1c value.
Measure: Least Squares Mean (Standard Error); unit: % change from baseline
Arm/Group | Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg | Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg | Treatment Naive: Empagliflozin 25 mg | Treatment Naive: Empagliflozin 10 mg | Treatment Naive: Linagliptin 5 mg
Number analyzed (Participants) | 134 | 135 | 133 | 132 | 133
% change from baseline | -1.08 (0.07) | -1.24 (0.07) | -0.95 (0.07) | -0.83 (0.07) | -0.67 (0.07)
Statistical Analysis 1: Comparison: Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg vs Treatment Naive: Empagliflozin 25 mg; Model for Week 24 includes baseline HbA1c (p<0.0001) as linear covariate(s) and baseline eGFR (MDRD) (p=0.8627), geographical region (p=0.0008), treatment (p<0.0001) as fixed effect(s); Test type: Superiority or Other; p = 0.1785, ANCOVA; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.33 to 0.06], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg vs Treatment Naive: Empagliflozin 10 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.41, 95% CI 2-sided [-0.61 to -0.21], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg vs Treatment Naive: Linagliptin 5 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Net) = -0.41, 95% CI 2-sided [-0.61 to -0.22], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg vs Treatment Naive: Linagliptin 5 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.57, 95% CI 2-sided [-0.76 to -0.37], Standard Error of Mean 0.10

6. Secondary Outcome: Change From Baseline in Body Weight for Treatment Naive Patients
Description: Change from baseline in body weight for Treatment Naive patients.
Time Frame: Baseline and 24 Weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kg change from baseline
Arm/Group | Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg | Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg | Treatment Naive: Empagliflozin 25 mg | Treatment Naive: Empagliflozin 10 mg | Treatment Naive: Linagliptin 5 mg
Number analyzed (Participants) | 134 | 135 | 133 | 132 | 133
kg change from baseline | -2.00 (0.36) | -2.74 (0.36) | -2.13 (0.36) | -2.27 (0.37) | -0.78 (0.36)
Statistical Analysis 1: Comparison: Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg vs Treatment Naive: Empagliflozin 25 mg; Model for Week 24 includes baseline weight (p<0.0001), baseline HbA1c (p=0.0023) as linear covariate(s) and baseline eGFR (MDRD) (p=0.0316), geographical region (p=0.0134), treatment (p=0.0031) as fixed effect(s); Test type: Superiority or Other; p = 0.8010, ANCOVA — Not an alpha protected test; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.88 to 1.14], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg vs Treatment Naive: Empagliflozin 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.3616, ANCOVA — Not an alpha protected test; Mean Difference (Net) = -0.47, 95% CI 2-sided [-1.48 to 0.54], Standard Error of Mean 0.51
Statistical Analysis 3: Comparison: Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg vs Treatment Naive: Linagliptin 5 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0178, ANCOVA; Mean Difference (Net) = -1.22, 95% CI 2-sided [-2.23 to -0.21], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg vs Treatment Naive: Linagliptin 5 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Net) = -1.96, 95% CI 2-sided [-2.97 to -0.95], Standard Error of Mean 0.51

7. Secondary Outcome: Occurrence of Treat to Target Efficacy Response for Metformin Background Patients
Description: Occurrence of the treat-to-target efficacy response for Metformin Background patients measured as HbA1c < 7.0% after 24 weeks of treatment for patients with HbA1c >=7.0% at baseline.
Time Frame: 24 Weeks
Population: Full Analysis Set (FAS) with non-completers considered failures (NCF). FAS- Metformin background patients randomised and treated who had a baseline (HbA1c>= 7% at baseline are included) and at least 1 on treatment HbA1c value with NCF approach, in which missing data due to premature discontinuation of a patient were considered as failure.
Measure: Number (95% Confidence Interval); unit: % of patients satisfying HbA1c <7.0%
Arm/Group | Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg | Metformin Background: Empagliflozin 25 mg | Metformin Background: Empagliflozin 10 mg | Metformin Background: Linagliptin 5 mg
Number analyzed (Participants) | 123 | 128 | 132 | 125 | 119
% of patients satisfying HbA1c <7.0% | 61.8 [52.6 to 70.4] | 57.8 [48.8 to 66.5] | 32.6 [24.7 to 41.3] | 28.0 [20.3 to 36.7] | 36.1 [27.5 to 45.4]
Statistical Analysis 1: Comparison: Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg vs Metformin Background: Empagliflozin 25 mg; Logistic regression includes treatment, baseline eGFR (MDRD), geographical region and baseline HbA1c; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.191, 95% CI 2-sided [2.319 to 7.573]
Statistical Analysis 2: Comparison: Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg vs Metformin Background: Empagliflozin 10 mg; Logistic regression includes treatment, baseline eGFR (MDRD), geographical region and baseline HbA1c; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.500, 95% CI 2-sided [2.474 to 8.184]
Statistical Analysis 3: Comparison: Metformin Background: Empagliflozin 25 mg/Linagliptin 5 mg vs Metformin Background: Linagliptin 5 mg; Logistic regression includes treatment, baseline eGFR (MDRD), geographical region and baseline HbA1c; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.495, 95% CI 2-sided [1.920 to 6.363]
Statistical Analysis 4: Comparison: Metformin Background: Empagliflozin 10 mg/Linagliptin 5 mg vs Metformin Background: Linagliptin 5 mg; Logistic regression includes treatment, baseline eGFR (MDRD), geographical region and baseline HbA1c; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 2.795, 95% CI 2-sided [1.562 to 5.001]

8. Secondary Outcome: Occurrence of Treat to Target Efficacy Response for Treatment Naive Patients
Description: Occurrence of the treat-to-target efficacy response for Treatment Naive patients measured as HbA1c < 7.0% after 24 weeks of treatment for patients with HbA1c >=7.0% at baseline.
Time Frame: 24 Weeks
Population: Full Analysis Set (FAS) with non-completers considered failures (NCF). FAS-treatment naive patients randomised and treated who had a baseline (HbA1c>= 7% at baseline are included) and at least 1 on treatment HbA1c value with NCF approach, in which missing data due to premature discontinuation of a patient were considered as failure.
Measure: Number (95% Confidence Interval); unit: % of patients satisfying HbA1c <7.0%
Arm/Group | Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg | Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg | Treatment Naive: Empagliflozin 25 mg | Treatment Naive: Empagliflozin 10 mg | Treatment Naive: Linagliptin 5 mg
Number analyzed (Participants) | 121 | 122 | 118 | 121 | 127
% of patients satisfying HbA1c <7.0% | 55.4 [46.1 to 64.4] | 62.3 [53.1 to 70.9] | 41.5 [32.5 to 51.0] | 38.8 [30.1 to 48.1] | 32.3 [24.3 to 41.2]
Statistical Analysis 1: Comparison: Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg vs Treatment Naive: Empagliflozin 25 mg; Logistic regression includes treatment, baseline eGFR (MDRD), geographical region and baseline HbA1c; Test type: Superiority or Other; p = 0.0224, Regression, Logistic; Odds Ratio (OR) = 1.893, 95% CI 2-sided [1.095 to 3.274]
Statistical Analysis 2: Comparison: Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg vs Treatment Naive: Empagliflozin 10 mg; Logistic regression includes treatment, baseline eGFR (MDRD), geographical region and baseline HbA1c; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.961, 95% CI 2-sided [1.697 to 5.169]
Statistical Analysis 3: Comparison: Treatment Naive: Empagliflozin 25 mg/Linagliptin 5 mg vs Treatment Naive: Linagliptin 5 mg; Logistic regression includes treatment, baseline eGFR (MDRD), geographical region and baseline HbA1c; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.065, 95% CI 2-sided [1.768 to 5.314]
Statistical Analysis 4: Comparison: Treament Naive: Empagliflozin 10 mg/Linagliptin 5 mg vs Treatment Naive: Linagliptin 5 mg; Logistic regression includes treatment, baseline eGFR (MDRD), geographical region and baseline HbA1c; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.303, 95% CI 2-sided [2.462 to 7.522]

ADVERSE EVENTS:
Time Frame: From first trial medication intake until 7 days after last drug intake during the 52-week study period
Description: One patient was randomized to treatment with Empa/Lina 25/5 but was treated with Empa 10 from the start of trial for 6 weeks. For efficacy, the patient was analyzed as randomized (Empa/Lina 25/5) and for safety the patient was analyzed as first medication taken (Empa 10).
Groups:
- Empagliflozin 25 mg/Linagliptin 5 mg: Test product: Empagliflozin/linagliptin FDC tablets dose: 25 mg/5 mg q.d. mode of admin.: Oral
- Empagliflozin 10 mg/Linagliptin 5 mg: Test product: Empagliflozin/linagliptin FDC tablets dose: 10 mg/5 mg q.d. mode of admin.: Oral
- Empagliflozin 25 mg: Reference therapy 1: Empagliflozin tablets dose: 25 mg q.d. mode of admin.: Oral
- Empagliflozin 10 mg: Reference therapy 1: Empagliflozin tablets dose: 10 mg q.d. mode of admin.: Oral
- Linagliptin 5 mg: Reference therapy 2: Linagliptin tablets dose: 5 mg q.d. mode of admin.: Oral
Arm/Group | Empagliflozin 25 mg/Linagliptin 5 mg | Empagliflozin 10 mg/Linagliptin 5 mg | Empagliflozin 25 mg | Empagliflozin 10 mg | Linagliptin 5 mg
Serious Adverse Events (participants affected / at risk) | 12/273 | 16/272 | 19/276 | 16/275 | 10/267
Other Adverse Events (participants affected / at risk) | 80/273 | 86/272 | 70/276 | 83/275 | 94/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 25 mg/Linagliptin 5 mg (N=273) | Empagliflozin 10 mg/Linagliptin 5 mg (N=272) | Empagliflozin 25 mg (N=276) | Empagliflozin 10 mg (N=275) | Linagliptin 5 mg (N=267)
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Encephalitis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Meningitis tuberculous (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 2 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Silent myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Chemical injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Finger amputation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 25 mg/Linagliptin 5 mg (N=273) | Empagliflozin 10 mg/Linagliptin 5 mg (N=272) | Empagliflozin 25 mg (N=276) | Empagliflozin 10 mg (N=275) | Linagliptin 5 mg (N=267)
Urinary tract infection (Infections and infestations) | 27 | 29 | 25 | 30 | 27
Nasopharyngitis (Infections and infestations) | 18 | 16 | 10 | 16 | 20
Upper respiratory tract infection (Infections and infestations) | 19 | 19 | 18 | 13 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 8 | 12 | 12 | 24
Headache (Nervous system disorders) | 16 | 15 | 13 | 19 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 14 | 13 | 10 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.